CLINICAL TRIAL: NCT02118909
Title: A Two-Part Study to Evaluate the Effect of CYP3A4 Inhibition (Itraconazole-Part 1) and CYP1A2 Inhibition (Ciprofloxacin - Part 2) on the Single-Dose Pharmacokinetics of Pracinostat in Healthy Nonsmoking Subjects
Brief Title: Evaluate the Effects of Itraconazole and Ciprofloxacin on Single-Dose PK of Pracinostat in Healthy Nonsmoking Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MEI-007
Record Dates: First submitted 2014-04-11; First posted 2014-04-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Healthy Volunteers; Non-smokers
MeSH Terms: interventions — SB939 compound; Itraconazole; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Pracinostat + Itraconazole) (Experimental): Single-dose pracinostat and itraconazole dosing every day for 8 days
  Interventions: Drug: Pracinostat; Drug: Ciprofloxacin
- Part 2 (Pracinostat + Ciprofloxacin) (Experimental): Single dose pracinostat and ciprofloxacin 2 times a day for 7 days
  Interventions: Drug: Pracinostat; Drug: Itraconazole

INTERVENTIONS:
Drug: Pracinostat
Drug: Itraconazole
  Arms: Part 2 (Pracinostat + Ciprofloxacin)
Drug: Ciprofloxacin
  Arms: Part 1 (Pracinostat + Itraconazole)

SUMMARY:
This study is designed as a 2-part, open-label study to assess the effect of pracinostat with itraconazole (part 1) and pracinostat with ciprofloxacin (part 2) on the bioavailability of pracinostat. Secondarily to evaluate the safety and tolerability of pracinostat administered with itraconazole or ciprofloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Continuous nonsmoker who has not used nicotine-containing products for at least 3 months prior to the first dose
* Body Mass Index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2 at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI.
* Female subjects must be of non-childbearing potential and must have undergone sterilization procedures at least 6 months prior to the first dose or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status.
* A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study medication.
* Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

* Subject is mentally or legally incapacitated or has significant emotional problems at the time of screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* History or presence of alcoholism or drug abuse within the past 2 years prior to screening.
* History or presence of hypersensitivity or idiosyncratic reaction to the study medication or related compounds.
* History of prolonged QT syndrome or require any current medications which may prolong QTc.
* History or presence of:

  * myasthenia gravis;
  * convulsions.
* Female subjects who are pregnant or lactating.
* Positive urine cotinine, drug and alcohol results at screening or check-in.
* Positive results at screening for HIV, HBsAg or HCV.
* Seated blood pressure is less than 90/40 mgHg or greater than 140/90 mmHg at screening.
* Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
* QTcF interval, is >430 msec (males) or >450 msec (females) or deemed clinical abnormal by the PI at screening or prior to dosing.
* Unable to refrain from or anticipates the use of:

  * Any drug, including prescription and non-prescription medications, tobacco, antacids, herbal remedies, or vitamin supplements beginning approximately 14 days prior to the first dose of study medication and throughout the study. Hormone replacement therapy will be allowed if postmenopausal females are on a stable treatment for at least 1 month prior to dosing on Day 1 of Period 1. Acetaminophen (up to 2 g per 24 hour period) may be permitted during the study.
  * Any drugs known to be significant inducers of CYP enzymes, including St. John's Wort, for 28 days prior to the first dose of study medication and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/pharmacodynamics interaction with study medication.
* Have been on a diet incompatible with the on-study diet, in the opinion of the PI, within the 28 days prior to the first dose of study medication(s), and throughout the study.
* Hemoglobin, platelet count or absolute neutrophils below the lower limit of normal at screening.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) above upper limit of normal at screening.
* Donation of blood or significant blood loss within 56 days prior to the first dose of study medication.
* Participation in another clinical trial within 28 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration Cmax in healthy nonsmoking subjects given a single-dose of pracinostat | pre-dose, 0.25, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours
  Plasma PK parameter Cmax to describe bioavailability of pracinostat

SECONDARY OUTCOMES:
Number of participants with Adverse Events as a measure of safety and tolerability of single-dose pracinostat when administered with itraconazole or with ciprofloxacin in healthy nonsmoking adult subjects. | 1 month
  Safety will be monitored through physical examinations, vital sign measurements, electrocardiograms, adverse events, and clinical laboratory tests.
Peak plasma PK concentration Area Under the Curve (AUC)AUC 0-t, AUC 0-inf in healthy nonsmoking subjects given a single dose of pracinostat | pre-dose, 0.25, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours
  Plasma PK parameter AUC 0-t, AUC 0-inf for pracinostat

CONTACTS AND LOCATIONS:
Overall Officials: Terry E O'Reilly, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States

REFERENCES:
- See also: Sponsor website — http://www.meipharma.com